CLINICAL TRIAL: NCT05328986
Title: Multi-center Assessment of Survivors for Kidney Disease After COVID-19
Brief Title: Kidney Disease After COVID-19
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: New Jersey Medical School (Other); University of Michigan (Other); Yale New Haven Health System Center for Healthcare Solutions (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Evren Azeloglu, Associate Professor of Medicine, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-20-01326; 1300143 (Other: Renalytix AI, Inc.)
Record Dates: First submitted 2022-04-13; First posted 2022-04-14 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: COVID-19; Acute Kidney Injury; Chronic Kidney Injury
MeSH Terms: conditions — COVID-19; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Collection of blood and urine samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID: Patients who have had a confirmed diagnosis of COVID-19.

SUMMARY:
To understand the long-term epidemiology, develop effective risk-prediction and stratification tools, and understand the pathobiology of kidney disease in COVID-19 survivors.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* Adults, age ≥18 years
* Confirmed diagnosis of COVID-19

Exclusion Criteria:

• No confirmed diagnosis of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 1753 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
estimated Glomerular Filtration Rate (eGFR) | yearly for 4 years after COVID exposure
  Kidneys filter blood by removing waste and extra water to make urine. The kidney's filtration rate, called the glomerular filtration rate (GFR), shows how well the kidneys are filtering. A normal GFR is 60 or higher.

SECONDARY OUTCOMES:
Urine Albumin-to-Creatinine Ratio (UACR) | yearly for 4 years after COVID exposure
  Albuminuria is present when UACR is greater than 30 mg/g and is a marker for chronic kidney disease. Albuminuria is used to diagnose and monitor kidney disease.
Urine protein/creatinine ratio (UPCR) | yearly for 4 years after COVID exposure
  Urine protein/creatinine ratio - Protein creatinine ratio in the urine quantifies the loss of the protein and helps in further evaluation of the kidney function. Normal ratio: < 0.20

CONTACTS AND LOCATIONS:
Overall Officials: Evren U. Azeloglu, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - Yale School of Medicine, New Haven, Connecticut
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - New Jersey Medical School - Rutgers University, Newark, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, CSR
Time Frame: Specify Other Time FrameData from this study may be requested from other researchers one year after the completion of the primary endpoint by contacting Dr. Evren Azeloglu.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Specify Other Mechanism
  1. Any research team who utilizes the data must propose a research question (independent and dependent variable) and post their plan for analysis on a COVID-19 database that is available.
  2. All teams need to abide by the requirement that data is analyzed within protected networks and that no data are downloaded or copied.
  3. Any data sharing will only occur with the approval with each site PI and only with appropriate regulatory approvals.
  Data will be deidentified.